CLINICAL TRIAL: NCT04115488
Title: Efficacy and Safety of the Biosimilar Natalizumab PB006 in Comparison to Tysabri® in Patients With Relapsing-Remitting Multiple Sclerosis (RRMS)
Brief Title: Efficacy and Safety of the Biosimilar Natalizumab PB006 in Comparison to Tysabri®
Acronym: Antelope
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polpharma Biologics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB006-03-01
Record Dates: First submitted 2019-09-10; First posted 2019-10-04 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PB006 (Experimental): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
  Interventions: Biological: Intravenous (IV) infusions
- Tysabri (Active Comparator): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006).
  Interventions: Biological: Intravenous (IV) infusions

INTERVENTIONS:
Biological: Intravenous (IV) infusions — Intravenous (IV) infusions of a dose of 300mg, every 4 weeks with a total of 12 doses

SUMMARY:
This is a multi-center, randomized, parallel arm, double-blind study with a total duration of subjects' participation of 48 weeks. Approximately 260 participants with relapsing-remitting multiple sclerosis will be randomized to receive 12 doses of either PB006 or EU-licensed Natalizumab.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter, double-blind, active-controlled, randomized, parallel-group study to assess the equivalence in efficacy and similarity in safety of biosimilar PB006 compared to Tysabri in patients with RRMS.

All eligible patients will be randomly assigned to one of two treatment groups in a 1:1 ratio, to receive a total of twelve intravenous (IV) infusion of either PB006 or Tysabri at a dose of 300 mg at each intravenous (IV) infusion administered with every single one intravenous (IV) infusion administered every 4 weeks of either PB006 or Tysabri at a dose of 300 mg starting at visit 1 (week 0) through visit 12 (week 44), for a total of 12 infusions. The End-of-Study Visit (visit 13, week 48) will be performed 4 weeks after the last infusion

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (age ≥18 to 60 years), with relapsing-remitting multiple sclerosis (RRMS) defined by the 2010 revised McDonald criteria
* At least 1 documented relapse within the previous year and either ≥1 GdE T1-weighted brain lesions or ≥9 T2-weighted brain lesions at Screening
* Kurtzke Expanded Disability Status Scale (EDSS) score from 0 to 5 (inclusive) at Screening

Exclusion Criteria:

* Manifestation of multiple sclerosis (MS) other than relapsing-remitting multiple sclerosis (RRMS)
* Relapse within the 30 days prior Screening and until administration of the first dose of study drug
* Prior treatment with natalizumab, alemtuzumab, ocrelizumab, daclizumab, rituximab, cladribine, or other B- and T-cell targeting therapies
* Prior total lymphoid irradiation or bone marrow or organ transplantation
* Patients with John Cunningham Virus (JCV) index >1.5 at Screening
* Past or current Progressive Multi-focal leukoencephalopathy (PML) diagnosis
* Severe renal function impairment as defined by serum creatinine values >120 micromol per litre

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Roth, Dr., Study Director — Polpharma Biologics S.A.
Locations (47):
- Belarus (6):
  - Grodno Regional Clinical Hospital, Grodno
  - Minsk City Clinical Hospital #5, Minsk
  - Republican Research and Development Center for Neurology and Neurosurgery, Minsk
  - Minsk Scientific and Practical Center of Surgery, Transplantology and Hematology, Minsk
  - Vitebsk Regional Diagnostic Center, Vitebsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Croatia (3):
  - Clinical Hospital Center Osijek, Clinic of Neurology, Osijek
  - Clinical Hospital Center Split, Clinic of Neurology, Split
  - University Hospital Centre Zagreb, Clinic of Neurology, Zagreb
- Georgia (6):
  - P. Sarajishvili Institute of Neurology, LTD, Tbilisi
  - LTD Saint Michael Archangel Multifunctional Clinical Hospital, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
  - LTD S.Khechinashvili University Hospital, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
- Moldova (2):
  - Institute for Emergency Medicine, Department of Neurology, Chisinau
  - National Institute of Neurology and Neurosurgery, Vascular Neurology Department, Chisinau
- Poland (6):
  - COPERNICUS Podmiot Leczniczy Sp. z o.o N. Copernicus Hospital, Department of Neurology, Gdansk, Pomeranian Voivodeship
  - Neuro-Medic, Katowice
  - Neurology Center Krzysztof Selmaj, Lodz
  - Provincial Specialist Hospital in Olsztyn, Department of Neurology, Olsztyn
  - MED-Polonia, Sp. z o.o. (LLC), Poznan
  - NeuroProtect Medical Center, Warsaw
- Serbia (4):
  - Clinical Center of Serbia, Clinic of Neurology, Belgrade
  - Clinical Hospital Center Zemun, Department of Neurology, Belgrade
  - Clinical Center Kragujevac, Clinic of Neurology, Kragujevac
  - Clinical Center of Vojvodina, Clinic of Neurology, Novi Sad
- Ukraine (20):
  - Cherkasy Regional Hospital of Cherkasy Oblast Council, Cherkasy
  - Dnipropetrovsk I.I. Mechnykov Regional Clinical Hospital, Dnipro
  - Ivano-Frankivsk City Clinical Hospital #1, Ivano-Frankivsk
  - Regional Clinical Hospital, Ivano-Frankivsk
  - City Clinical Hospital #7, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology, Kharkiv
  - Kharkiv Railway Clinical Hospital, Kharkiv
  - Kyiv City Clinical Hospital, Kyiv
  - Medical Center of First Private Clinic, Kyiv
  - National Research Center for Radiation Medicine, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv
  - Lviv City Clinical Hospital #5, Lviv
  - Center for Reconstructive and Restorative Medicine (University Clinic), Odesa
  - Sklifosovskyi Regional Clinical Hospital, Poltava
  - Ternopil Regional Clinical Psychonevrological Hospital, Ternopil
  - Vinnytsia O.I. Yushchenko Regional Psychoneurology Hospital, Vinnytsia
  - Clinical Hospital No. 9 under Zaporizhia City Council, Zaporizhia
  - City Clinical Hospital #2, Zaporizhzhya
  - Zaporizhia Regional Clinical Hospital, Zaporizhzhya
  - O.F. Herbachevskyi Regional Clinical Hospital, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hemmer B, Wiendl H, Roth K, Wessels H, Hofler J, Hornuss C, Liedert B, Selmaj K. Efficacy and Safety of Proposed Biosimilar Natalizumab (PB006) in Patients With Relapsing-Remitting Multiple Sclerosis: The Antelope Phase 3 Randomized Clinical Trial. JAMA Neurol. 2023 Mar 1;80(3):298-307. doi: 10.1001/jamaneurol.2022.5007. PMID 36689214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3 multicenter, double-blind, active-controlled, randomized, parallel-group study to assess the similarity in efficacy, safety, and immunogenicity of biosimilar natalizumab PB006 compared to European Union-approved Tysabri in patients with Relapsing-remitting multiple sclerosis (RRMS).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. One subject withdrew consent before receiving study drug and was not included in the results.
Period: Overall Study
Arm/Group | PB006 | Tysabri
Started | 131 | 133
Patients Re-randomized and Switched From Tysabri to PB006 at Week 24. | 0 | 30
Patients Continuing on Tysabri Following the Re-randomization at Week 24. | 0 | 95
Completed | 117 | 122
Not Completed | 14 | 11
Not completed — Adverse Event | 8 | 4
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Investigator/ Sponsor Decision | 2 | 0
Not completed — Patient 's location change | 1 | 0
Not completed — Due to COVID-19 restrictions at site | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) Population includes all patients who were randomized and have received at least one infusion of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PB006 | Tysabri | Total
Number analyzed (Participants) | 131 | 133 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (9.05) | 36.6 (9.73) | 36.7 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 78 | 162
  Male | 47 | 55 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 133 | 264
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 131 | 133 | 264
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of New Active Lesions Over 24 Weeks
Description: Cumulative number of new active lesions over 24 weeks, calculated as the sum of all new gadolinium-enhancing (GdE) T1-weighted and new/enlarging T2-weighted lesion. Assessment was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted and T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center.
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20 and 24.
Population: Per-Protocol: patients who completed the 24-week treatment period without major protocol deviations that may have influenced the analysis of the primary endpoint and for whom sufficient post-baseline MRI data were available (baseline, Week 24 and at least 1/3 MRI visits). Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switched or not. Subjects with non-missing endpoints in the analysis.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- PB006 (Per-Protocol): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
- Tysabri (Per-Protocol): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006).
- PB006 (Safety-Switch): Patients with relapsing-remitting multiple sclerosis (RRMS) received IV infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
- Tysabri Switched to PB006 at Week 24 (Safety-Switch): Patients with relapsing-remitting multiple sclerosis (RRMS) received IV infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006). This arm concerns patients who started on Tysabri and continued on PB006 following the re-randomization at week 24.
- Tysabri Continued at Week 24 (Safety-Switch): Patients with relapsing-remitting multiple sclerosis (RRMS) received IV infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. This arm concerns patients who started on Tysabri and continued on Tysabri following the re-randomization at week 24.
Arm/Group | PB006 (Per-Protocol) | Tysabri (Per-Protocol) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 111 | 118 | 122 | 30 | 95
lesions | 1.4 (3.73) | 1.9 (3.97) | 1.4 (3.65) | 2.1 (3.78) | 1.9 (4.09)
Statistical Analysis 1: Comparison: PB006 (Per-Protocol) vs Tysabri (Per-Protocol); Test type: Equivalence — Data was analyzed using a negative binomial model with a logarithmic link function and fixed effects for the treatment group and stratification factors. Equivalence was tested based 95% confidence interval; Exponentiated Difference = 0.17, 95% CI 2-sided [-0.613 to 0.944], Standard Error of Mean 0.397 — Difference calculated as Tysabri minus PB006

2. Secondary Outcome: Cumulative Number of New Active Lesions Over 48 Weeks
Description: Cumulative number of new active lesions over 48 weeks, calculated as the sum of all new gadolinium-enhancing (GdE) T1-weighted and new/enlarging T2-weighted lesion. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions and T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent was administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switched or not. Subjects with non-missing endpoints in the analysis.
  Tysabri (FAS): Patients who switch from Tysabri to PB006 are excluded.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- PB006 (Full Analysis Set): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
- Tysabri (Full Analysis Set): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006).
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 122 | 96 | 119 | 29 | 95
lesions | 1.5 (3.72) | 2.3 (5.68) | 1.5 (3.75) | 2.1 (3.82) | 2.3 (5.70)

3. Secondary Outcome: Cumulative Number of New GdE T1-weighted Lesions Over 24 Weeks
Description: Cumulative number of new GdE T1-weighted lesions over 24 weeks, calculated as the sum of all new gadolinium-enhancing (GdE) T1-weighted. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20 and 24.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switched or not. Subjects with non-missing endpoints in the analysis.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 126 | 127 | 122 | 30 | 95
lesions | 0.3 (1.01) | 0.4 (1.25) | 0.3 (1.02) | 0.4 (0.81) | 0.4 (1.37)

4. Secondary Outcome: Cumulative Number of New GdE T1-weighted Lesions Over 48 Weeks
Description: Cumulative number of new GdE T1-weighted lesions over 48 weeks, calculated as the sum of all new gadolinium-enhancing (GdE) T1-weighted. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: The Full Analysis Set (FAS) population: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch (SSW) Population: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 122 | 96 | 119 | 29 | 95
lesions | 0.3 (1.02) | 0.4 (1.39) | 0.3 (1.03) | 0.4 (0.82) | 0.4 (1.40)

5. Secondary Outcome: Number of Patients Without New GdE T1-weighted Lesions Over 24 Weeks
Description: Number of patients without new GdE T1-weighted lesions over 24 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20 and 24.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not.
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 133 | 122 | 30 | 95
Participants | 109 | 105 | 105 | 23 | 80

6. Secondary Outcome: Number of Patients Without New GdE T1-weighted Lesions Over 48 Weeks
Description: Number of patients without new GdE T1-weighted lesions over 48 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
  Tysabri (FAS): Patients who switch from Tysabri to PB006 are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 103 | 122 | 30 | 95
Participants | 105 | 80 | 102 | 22 | 79

7. Secondary Outcome: Cumulative Number of New/Enlarging T2-weighted Lesions Over 24 Weeks
Description: Cumulative number of new/enlarging T2-weighted lesions over 24 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center.
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20 and 24.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 126 | 127 | 122 | 30 | 95
lesions | 1.5 (3.79) | 2.0 (4.12) | 1.5 (3.83) | 2.2 (3.84) | 2.0 (4.25)

8. Secondary Outcome: Cumulative Number of New/Enlarging T2-weighted Lesions Over 48 Weeks
Description: Cumulative number of new/enlarging T2-weighted lesions over 48 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center.
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 122 | 96 | 119 | 29 | 95
lesions | 1.6 (3.09) | 2.4 (5.79) | 1.6 (3.93) | 2.2 (3.89) | 2.5 (5.81)

9. Secondary Outcome: Number of Persistent Lesions After 24 Weeks
Description: Number of persistent lesions after 24 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions and T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20 and 24.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch : treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 126 | 127 | 122 | 30 | 95
lesions | 0.5 (2.46) | 0.4 (2.92) | 0.5 (2.49) | 0.1 (0.31) | 0.6 (3.37)

10. Secondary Outcome: Number of Persistent Lesions After 48 Weeks
Description: Number of persistent lesions after 48 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of GdE T1-weighted lesions and T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center. A macrocyclic Gd-based contrast agent (gadobutrol, gadoteric acid, or gadoteridol) was to be administered as an Intravenous infusion of 0.1 Millimole per kilogram [mmol/kg].
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 122 | 96 | 119 | 29 | 95
lesions | 0.5 (2.55) | 0.6 (3.35) | 0.5 (2.58) | 0.1 (0.26) | 0.6 (3.37)

11. Secondary Outcome: Annualized Relapse Rate After 24 Weeks
Description: Annualized relapse rate after 24 weeks. Relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality had to be present for at least 24 hours and have occurred in the absence of fever or infection. Annualized relapse rate: A: Number of medically confirmed relapses overall. B: Duration of follow-up time overall, where follow-up time was defined as: (last day of follow-up - day of randomization + 1) / 365.25. The ratio of relapses per patient-year: A/B. Annualized Relapse Rate was calculated across the entire group.
Time Frame: Up to 24 weeks.
Population: Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not.
Measure: Number; unit: Relapses per patient-year
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 133 | 122 | 30 | 95
Relapses per patient-year | 0.206 | 0.152 | 0.194 | 0.143 | 0.114

12. Secondary Outcome: Annualized Relapse Rate After 48 Weeks
Description: Annualized relapse rate after 48 weeks. Relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality had to be present for at least 24 hours and have occurred in the absence of fever or infection. Annualized relapse rate: A: Number of medically confirmed relapses overall. B: Duration of follow-up time overall, where follow-up time was defined as: (last day of follow-up - day of randomization + 1) / 365.25. The ratio of relapses per patient-year: A/B. Annualized Relapse Rate was calculated across the entire group.
Time Frame: Up to 48 weeks.
Population: Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
  Tysabri (FAS): Patients who switch from Tysabri to PB006 are excluded.
Measure: Number; unit: Relapses per patient-year
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 103 | 122 | 30 | 95
Relapses per patient-year | 0.174 | 0.133 | 0.168 | 0.146 | 0.113

13. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) After 24 Weeks
Description: Change from baseline in Expanded Disability Status Scale (EDSS) after 24 weeks. The Kurtzke EDSS, commonly used to evaluate the degree of neurologic impairment in multiple sclerosis (MS), is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. Based on a standard neurological examination, the 7 functional systems (plus "other") are rated. These ratings are then used in conjunction with observations and information concerning gait and use of assistive devices to rate the EDSS. EDSS ratings were performed by independent examining neurologists. After re-randomization, Week 24 is considered baseline.
Time Frame: Baseline and week 24.
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 122 | 125
score on a scale | -0.03 (0.211) | 0.00 (0.354)

14. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) After 48 Weeks
Description: Change from baseline in Expanded Disability Status Scale (EDSS) after 48 weeks. The Kurtzke EDSS, commonly used to evaluate the degree of neurologic impairment in MS, is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. Based on a standard neurological examination, the 7 functional systems (plus "other") are rated. These ratings are then used in conjunction with observations and information concerning gait and use of assistive devices to rate the EDSS. EDSS ratings were performed by independent examining neurologists.
Time Frame: FAS: Baseline (week 0) and week 48. SSW: Baseline (week 24) and week 48.
Population: Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
  Tysabri (FAS): Patients who switch from Tysabri to PB006 are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 117 | 93 | 117 | 29 | 93
score on a scale | -0.14 (0.536) | -0.05 (0.443) | -0.10 (0.498) | -0.03 (0.325) | -0.02 (0.312)

15. Secondary Outcome: Percentage of Subjects With Anti-drug (Natalizumab) Antibodies (ADA) and Persistent Antibodies After 24 Weeks
Description: Percentage of subjects with anti-drug (natalizumab) antibodies (ADA) and persistent antibodies after 24 weeks. A positive ADA patient was defined as a patient who had at least 1 positive ADA result in any post-baseline sample. A persistently positive ADA patient was defined as a patient with confirmed positive ADAs in 2 or more consecutive positive ADA samples at post-dose visits.
Time Frame: Up to 24 weeks.
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF). Patients in this group were analyzed as treated. Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
Measure: Number; unit: Percentage of subjects
Groups:
- PB006 (Safety): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
- Tysabri (Safety): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006).
Arm/Group | PB006 (Safety) | Tysabri (Safety) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 122 | 125 | 122 | 30 | 95
Percentage of subjects
  Persistently positive (confirmed) | 28.7 | 27.2 | 28.7 | 43.3 | 22.1
  Positive, confirmed | 30.3 | 29.6 | 30.3 | 43.3 | 25.3

16. Secondary Outcome: Percentage of Subjects With Anti-drug (Natalizumab) Antibodies (ADA) and Persistent Antibodies After 48 Weeks
Description: Percentage of subjects with anti-drug (natalizumab) antibodies (ADA) and persistent antibodies after 48 weeks. A positive ADA patient was defined as a patient who had at least 1 positive ADA result in any post-baseline sample. A persistently positive ADA patient was defined as a patient with confirmed positive ADAs in 2 or more consecutive positive ADA samples at post-dose visits.
Time Frame: Up to 48 weeks.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | PB006 (Safety) | Tysabri (Safety) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 115 | 121 | 115 | 28 | 93
Percentage of subjects
  Persistently positive (confirmed) | 10.4 | 11.6 | 10.4 | 17.9 | 9.7
  Positive, confirmed) | 11.3 | 11.6 | 11.3 | 17.9 | 9.7

17. Secondary Outcome: Percentage of Subjects With Neutralizing Antibodies After 24 Weeks
Description: Percentage of subjects with positive (transient and persistent) neutralizing antibodies after 24 weeks.
Time Frame: Up to 24 weeks.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | PB006 (Safety) | Tysabri (Safety) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 37 | 37 | 37 | 13 | 24
Percentage of subjects | 67.6 | 64.9 | 67.6 | 61.5 | 66.7

18. Secondary Outcome: Percentage of Subjects With Neutralizing Antibodies After 48 Weeks
Description: Percentage of subjects with positive (transient and persistent) neutralizing antibodies after 48 weeks.
Time Frame: Up to 48 weeks.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | PB006 (Safety) | Tysabri (Safety) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 13 | 14 | 13 | 5 | 9
Percentage of subjects | 61.5 | 50.0 | 61.5 | 60.0 | 44.4

19. Secondary Outcome: Number of Subjects With Any Treatment-Emergent Adverse Event (TEAE) or Any Treatment-Emergent Serious Adverse Event (SAE) After 24 Weeks
Description: Number of subjects with any Treatment-Emergent Adverse Event (TEAE) or any Treatment-Emergent Serious Adverse Event (SAE) after 24 weeks.
Time Frame: Up to week 24
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF). Patients in this group were analyzed as treated.
Measure: Number; unit: participants
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 131 | 133
participants
  TEAE | 62 | 64
  Treatment-emergent SAE | 1 | 0

20. Secondary Outcome: Number of Subjects With Any Treatment-Emergent Adverse Event (TEAE) or Any Treatment-Emergent Serious Adverse Event (SAE) After 48 Weeks
Description: Number of subjects with any Treatment-Emergent Adverse Event (TEAE) or any Treatment-Emergent Serious Adverse Event (SAE) after 48 weeks.
Time Frame: Up to 48 weeks.
Population: as for outcome 19
Measure: Number; unit: participants
Groups:
- Tysabri Switched to PB006 at Week 24 (Safety): Patients with relapsing-remitting multiple sclerosis (RRMS) received IV infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006). This arm concerns patients who started on Tysabri and continued on PB006 following the re-randomization at week 24.
- Tysabri Continued at Week 24 (Safety): Patients with relapsing-remitting multiple sclerosis (RRMS) received IV infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. This arm concerns patients who started on Tysabri and continued on Tysabri following the re-randomization at week 24.
Arm/Group | PB006 (Safety) | Tysabri Switched to PB006 at Week 24 (Safety) | Tysabri Continued at Week 24 (Safety)
Number analyzed (Participants) | 131 | 30 | 103
participants
  TEAE | 85 | 22 | 71
  Treatment-emergent SAE | 3 | 0 | 2

21. Secondary Outcome: Natalizumab Trough Concentration (Ctrough) Over Time, Week 8
Description: Natalizumab trough concentration (Ctrough) over time, week 8. Serum samples were collected prior to treatment. Sample was taken prior to treatment for each patient.
Time Frame: Week 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 118 | 125
Nanograms per milliliter (ng/mL) | 26804.75 (12949.541) | 25010.49 (12557.895)

22. Secondary Outcome: Natalizumab Trough Concentration (Ctrough) Over Time, Week 16
Description: Natalizumab trough concentration (Ctrough) over time, week 16. Serum samples were collected prior to treatment. Sample was taken prior to treatment for each patient.
Time Frame: Week 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 117 | 122
Nanograms per milliliter (ng/mL) | 33872.92 (18151.190) | 32543.28 (14636.925)

23. Secondary Outcome: Natalizumab Trough Concentration (Ctrough) Over Time, Week 24
Description: Natalizumab trough concentration (Ctrough) over time, week 24. Serum samples were collected prior to treatment. Sample was taken prior to treatment for each patient.
Time Frame: Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 117 | 121
Nanograms per milliliter (ng/mL) | 36853.93 (15292.389) | 35617.65 (16049.669)

24. Secondary Outcome: Natalizumab Trough Concentration (Ctrough) Over Time, Week 32
Description: Natalizumab trough concentration (Ctrough) over time, week 32. Serum samples were collected prior to treatment. Sample was taken prior to treatment for each patient.
Time Frame: Week 32
Population: The Full Analysis Set: patients who were randomized and have received at least one (complete or partial) infusion of the study drug. Only subjects with non-missing endpoints were included in the analysis. For this outcome measure, only participants who remain in the same treatment group through study period were included.
  Only patients who stayed on their randomized treatment were included in the endpoint, patients who switch from Tysabri to PB006 were excluded.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 115 | 94
Nanograms per milliliter (ng/mL) | 37450.04 (16877.010) | 36865.81 (19756.050)

25. Secondary Outcome: Natalizumab Trough Concentration (Ctrough) Over Time, Week 48
Description: Natalizumab trough concentration (Ctrough) over time, week 48. Serum samples were collected prior to treatment. Sample was taken prior to treatment for each patient.
Time Frame: Week 48
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 110 | 91
Nanograms per milliliter (ng/mL) | 39097.58 (16801.710) | 38432.86 (16495.407)

26. Secondary Outcome: Number of Patients Without New/Enlarging T2-weighted Lesions Over 24 Weeks
Description: Number of patients without new/enlarging T2-weighted lesions over 24 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center.
Time Frame: Week 0 (baseline), week 8, 16, 20 and 24.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 133 | 122 | 30 | 95
Participants | 75 | 72 | 72 | 18 | 52

27. Secondary Outcome: Number of Patients Without New/Enlarging T2-weighted Lesions Over 48 Weeks
Description: Number of patients without new/enlarging T2-weighted lesions over 48 weeks. Assessment of lesions was performed using Magnetic Resonance Imaging (MRI). Identification of T2-weighted lesions was done by a trained and certified radiology reviewer according to standard procedures at the MRI central reading center.
Time Frame: Scans performed at week 0 (baseline), week 8, 16, 20, 24 and 48.
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Full Analysis Set) | Tysabri (Full Analysis Set) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 131 | 103 | 122 | 30 | 95
Participants | 71 | 52 | 69 | 17 | 51

28. Secondary Outcome: Number of Patients With Abnormal Clinical Laboratory Tests at Week 24
Description: Number of patients with abnormal clinical laboratory tests at week 24.
Time Frame: At week 24.
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF).
Measure: Count of Participants; unit: Participants
Groups:
- PB006 (Safety Population): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions.
- Tysabri (Safety Population): Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of Tysabri at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. At Week 24, patients in the Tysabri group were re-randomized through a re-randomization step. Patients re-randomized and switched from Tysabri to PB006 at Week 24 still received a total of 12 infusions (6 infusions of Tysabri and 6 infusions of PB006).
Arm/Group | PB006 (Safety Population) | Tysabri (Safety Population)
Number analyzed (Participants) | 122 | 125
Participants | 116 | 114

29. Secondary Outcome: Number of Patients With Abnormal Clinical Laboratory Tests at Week 48
Description: Number of patients with abnormal clinical laboratory tests at week 48.
Time Frame: At week 48.
Population: Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switched or not.
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 117 | 29 | 93
Participants | 108 | 26 | 88

30. Secondary Outcome: Number of Patients With Abnormal Findings in Physical Examination at Week 24
Description: Number of patients with abnormal findings in physical examination at week 24.
Time Frame: Week 24.
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 122 | 125
Participants | 10 | 12

31. Secondary Outcome: Number of Patients With Abnormal Findings in Physical Examination at Week 48
Description: Number of patients with abnormal findings in physical examination at week 48.
Time Frame: End of study (week 48).
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF).
  Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switched or not.
Measure: Count of Participants; unit: Participants
Arm/Group | PB006 (Safety) | Tysabri (Safety) | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 117 | 122 | 117 | 29 | 93
Participants | 11 | 10 | 11 | 3 | 7

32. Secondary Outcome: Change From Baseline in Blood Pressure at Week 24
Description: Change from baseline in diastolic and systolic blood Pressure at week 24.
Time Frame: At baseline and week 24.
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF). Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 122 | 125
Millimeter of mercury (mmHg)
  Diastolic Blood Pressure | -2.2 (7.30) | -0.6 (7.35)
  Systolic Blood Pressure | -1.0 (9.76) | -1.5 (11.33)

33. Secondary Outcome: Change From Baseline in Blood Pressure at Week 48
Description: Change from baseline in diastolic and systolic blood Pressure at week 48.
Time Frame: At baseline and end of study (week 48).
Population: Safety-Switch Population: Patients who were included in the SAF and received at least 1 infusion of the study drug after the timepoint of re-randomization, independent of whether they switched or not, were included in the Safety-Switch Population (SSW). Patients in this group were analyzed as treated after re-randomization, also considering treatment before re-randomization.
  Tysabri (SSW): Patients who switch from Tysabri to PB006 are excluded.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 117 | 29 | 93
Millimeter of mercury (mmHg)
  Diastolic Blood Pressure | 1.0 (7.58) | 1.8 (8.16) | 0.8 (7.68)
  Systolic Blood Pressure | 1.7 (8.67) | 2.4 (12.38) | 3.0 (10.18)

34. Secondary Outcome: Change From Baseline in Heart Rate at Week 24
Description: Change from baseline in heart rate at week 24.
Time Frame: At baseline and week 24.
Population: Safety Population: Patients who received at least 1 (complete or partial) infusion of the study drug were included in the Safety Population (SAF). Patients in this group were analyzed as treated. Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | PB006 | Tysabri
Number analyzed (Participants) | 122 | 125
beats/minute | -0.4 (9.05) | -1.4 (9.10)

35. Secondary Outcome: Change From Baseline in Heart Rate at Week 48
Description: Change from baseline in heart rate at week 48.
Time Frame: At baseline and end of study (week 48).
Population: Safety-Switch: treated patients who received at least one infusion of the study drug after the time point of re-randomization, independent of whether they switch or not. Only subjects with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | PB006 (Safety-Switch) | Tysabri Switched to PB006 at Week 24 (Safety-Switch) | Tysabri Continued at Week 24 (Safety-Switch)
Number analyzed (Participants) | 117 | 29 | 93
beats/minute | 0.8 (7.07) | 1.7 (10.53) | 1.1 (9.66)

ADVERSE EVENTS:
Time Frame: From first infusion till the last + 4 weeks, up to 48 weeks. Deaths (all causes): From first infusion till the last (at Week 44) + 24 ± 2 weeks, up to 68 ± 2 weeks.
Description: Patients participating in this study who receive at least one (complete or partial) infusion of the study drug were included in the Safety Population (SAF).
Groups:
- PB006: Patients with relapsing-remitting multiple sclerosis (RRMS) received intravenous (IV) infusions every 4 weeks of PB006 at a dose of 300 milligram (mg) starting at Visit 1 (Week 0) through Visit 12 (Week 44), for a total of 12 infusions. This arm includes patients who switched from Tysabri to PB006 during the re-randomization step at week 24.
Arm/Group | PB006 | Tysabri
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/133
Serious Adverse Events (participants affected / at risk) | 3/161 | 2/133
Other Adverse Events (participants affected / at risk) | 100/161 | 93/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PB006 (N=161) | Tysabri (N=133)
Hypotension (Vascular disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PB006 (N=161) | Tysabri (N=133)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Asthenia (General disorders) | 5 | 2
Fatigue (General disorders) | 5 | 1
Pyrexia (General disorders) | 1 | 4
Hyperthermia (General disorders) | 2 | 1
Feeling hot (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 1
Discomfort (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 4 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 1 | 0
Weight decreased (Investigations) | 2 | 4
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 1 | 2
C-reactive protein increased (Investigations) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Bilirubin conjugated increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Scar (Investigations) | 1 | 0
Thermal burn (Investigations) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Headache (Nervous system disorders) | 27 | 23
Dizziness (Nervous system disorders) | 3 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 2 | 1
Tension headache (Nervous system disorders) | 2 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Head titubation (Nervous system disorders) | 0 | 1
Hyposmia (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Skin and subcutaneous tissue disorders) | 0 | 1
Nephroptosis (Skin and subcutaneous tissue disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 14 | 13
COVID-19 (Infections and infestations) | 14 | 10
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Pharyngitis (Infections and infestations) | 1 | 4
Respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 3
Cystitis (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infected fistula (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyoderma streptococcal (Infections and infestations) | 1 | 1
Tinea versicolour (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04115488/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04115488/SAP_001.pdf